CLINICAL TRIAL: NCT03106714
Title: Study on the Persistence of Zika Virus (ZIKV) in Body Fluids of Patients With ZIKV Infection in Brazil
Acronym: ZikaBra
Status: Completed | Type: Observational
Sponsor: Oswaldo Cruz Foundation (Other)
Collaborators: World Health Organization (Other); Ministry of Health, Brazil (Other Government); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); Wellcome Trust (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Guilherme Amaral Calvet, MD, PhD, Oswaldo Cruz Foundation
Other Study IDs: ERC.0002786; 62518016.6.1001.0008 (Other: Brazil National Commission for Research Ethics); R21AI139777 (NIH); TSA1-2017/720873-0 (Other Grant/Funding Number: World Health Organization); TSA2-2017/731359-0 (Other Grant/Funding Number: World Health Organization); 206522/Z/17/Z (Other Grant/Funding Number: Wellcome Trust); Convênio 837059/2016 (Other Grant/Funding Number: Brazilian Ministry of Health); W81XWH-18-2-0040 (Other Grant/Funding Number: Henry M. Jackson Foundation)
Record Dates: First submitted 2017-04-03; First posted 2017-04-10 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Zika Virus
Keywords: persistence; body fluids
MeSH Terms: conditions — Zika Virus Infection | interventions — COVID-19 Nucleic Acid Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples with DNA: whole blood and PBMC Also collected and stored: serum, semen, saliva, crevicular fluid, urine, vaginal secretions, menstrual blood, rectal swab, tears, sweat, and breast milk
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Detectable RT-PCR ZIKV: Men and women aged 18 years and above with diagnosis of ZIKV infection
  Interventions: Diagnostic Test: RT-PCR

INTERVENTIONS:
Diagnostic Test: RT-PCR — Persistence of detectable Zika virus (by RT-PCR test) in all selected body fluids

SUMMARY:
The Zika infection is a viral disease that is transmitted to humans by the same mosquito that transmits Dengue and Chikungunya fever. The Zika virus has been found in various body fluids such as urine, blood and semen, but we do not know how long it persists in these fluids. For example, parts of the virus were reported to persist in semen after six months of the onset of symptoms, but we do not know if the virus can stay longer. In this way, we want to investigate how long the Zika virus can be found in other secretions besides blood and urine.

Study Hypothesis: ZIKV can be shed in human body fluids long after the time of the acute infection. Persistence of ZIKV in different body fluids may vary due to the influence of circulating specific ZIKV IgM and IgG, as well as host and environmental factors.

DETAILED DESCRIPTION:
Little is known about Zika virus (ZIKV) biology and its pathogenesis in humans. ZIKV has been detected in blood, urine, semen, cerebral spinal fluid, saliva, amniotic fluid, and breast milk. In most ZIKV infected individuals, the virus is detected in the blood from a several days to one week after the onset of symptoms and has also been found to persist longer in urine and semen. Without a more granular understanding of the kinetics of ZIKV infection across biologic compartments it will be difficult to devise rational measures to prevent the transmission of the virus.

This will be an observational cohort study of men and women, aged 18 years and above, including symptomatic participants with positive reverse transcriptase-polymerase chain reaction (RT-PCR) test in blood and/or urine and their symptomatic or asymptomatic household/sexual contacts with positive RT-PCR in blood and/or urine. Specimens to be collected at pre-established intervals and tested for ZIKV RNA by RT-PCR are blood, semen, vaginal secretions, oral fluid (saliva and crevicular fluid), tears, sweat, urine, rectal swab, menstrual blood and breast milk (if applicable). Participants will be recruited from collaborating clinics in selected locations with high population density, high circulation of the virus, strong community network, and serviced by laboratory facilities with capacity to perform the necessary tests.

All participants will be followed up for 12 months, to assess detectability at longer time intervals, reactivation or reinfection. Analyses of antibody response, including circulating immunoglobulins M and G (IgM and IgG), will be performed in parallel to RT-PCR tests. Plaque reduction neutralization test will be performed in specimens of participants who are found to be simultaneously positive for ZIKV and dengue.

Specific analysis will be performed to determine if socio-demographic characteristics, comorbidities and co-infections influence the persistence of the virus in the body fluids.

ELIGIBILITY:
Index Case - Enrolment Inclusion criteria

* RT-PCR test positive for ZIKV in blood and/or urine specimens
* Having given consent to provide all body fluid collection, as per protocol

Exclusion criteria RT-PCR test negative for ZIKV in blood and/or urine specimens

Household contacts enrollment (or sexual contacts if index case lives alone) Inclusion criteria

* As per index case Exclusion criteria
* As per index case

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective observational cohort study. After signing a screening consent, male and female potential study participants presenting rash compatible with ZIKV infection in collaborating clinics will be tested for the presence of ZIKV in blood and urine. The following day, after providing informed consent for enrolment, those found to be RT-PCR positive for ZIKV infection, fulfilling all inclusion criteria will be enrolled and subject of regular collection of body fluids over a period of 12 months according to a pre-established schedule. Household/sexual contacts will be screened at the reference centers where the index case was diagnosed or if preferable at their household, and recruited following the same criteria. The standard care will be provided to all participants.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Persistence and duration of ZIKV | 12 months of follow-up after ZIKV infection diagnosis
  Persistence and duration of ZIKV in each body fluid in infected symptomatic and asymptomatic participants.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie JN Broutet, MD, PhD, Study Chair — Department of Reproductive Health and Research World Health Organization; Ana Maria B de Filippis, PhD, Principal Investigator — Oswaldo Cruz Foundation (Flavivirus Diagnostic and Reference Laboratory- Rio de Janeiro); Guilherme A Calvet, MD,PhD, Principal Investigator — Oswaldo Cruz Foundation (Evandro Chagas National Institute of Infectious Diseases- Rio de Janeiro); Rafael FO França, PhD, Principal Investigator — Oswaldo Cruz Foundation (Research Centre Aggeu Magalhães- Recife); Marcus VG Lacerda, MD,PhD, Principal Investigator — Tropical Medicine Foundation, Manaus
Locations (3):
- Brazil (3):
  - Tropical Medicine Foundation, Manaus, Amazonas
  - Research Centre Aggeu Magalhães, Oswaldo Cruz Foundation, Recife, Pernambuco
  - Evandro Chagas National Institute of Infectious Diseases - Oswaldo Cruz Foundation, Rio de Janeiro

REFERENCES:
- [Background] Calvet GA, Kara EO, Giozza SP, Botto-Menezes CHA, Gaillard P, de Oliveira Franca RF, de Lacerda MVG, da Costa Castilho M, Brasil P, de Sequeira PC, de Mello MB, Bermudez XPD, Modjarrad K, Meurant R, Landoulsi S, Benzaken AS, de Filippis AMB, Broutet NJN; ZIKABRA Study Team. Study on the persistence of Zika virus (ZIKV) in body fluids of patients with ZIKV infection in Brazil. BMC Infect Dis. 2018 Jan 22;18(1):49. doi: 10.1186/s12879-018-2965-4. PMID 29357841
- [Result] Menezes-Neto A, Castilho MDC, Calvet GA, Kara EO, Botto-Menezes CHA, Lacerda MVG, Pereira GFM, Giozza SP, Bermudez XPD, Lima NS, Modjarrad K, Broutet N, de Filippis AMB, Franca RFO; Study Team ZIKABRA. Zika virus RNA excretion in sweat with concomitant detection in other body fluid specimens. Mem Inst Oswaldo Cruz. 2021 Jan 25;115:e200339. doi: 10.1590/0074-02760200339. eCollection 2021. PMID 33503145
- [Result] Calvet GA, Kara EO, Landoulsi S, Habib N, Botto-Menezes CHA, Franca RFO, Neto AM, Castilho MDC, Fernandes TJ, Pereira GF, Giozza SP, Bermudez XPD, Modjarrad K, Lima N, Brasil P, de Lacerda MVG, de Filippis AMB, Broutet NJN; ZIKABRA Study Team. Cohort profile: Study on Zika virus infection in Brazil (ZIKABRA study). PLoS One. 2021 Jan 5;16(1):e0244981. doi: 10.1371/journal.pone.0244981. eCollection 2021. PMID 33400705
- [Result] Botto-Menezes CHA, Neto AM, Calvet GA, Kara EO, Lacerda MVG, Castilho MDC, Stroher U, Antunes de Brito CA, Modjarrad K, Broutet N, Brasil P, Bispo de Filippis AM, Franca RFO; ZIKABRA Study Team. Zika Virus in Rectal Swab Samples. Emerg Infect Dis. 2019 May;25(5):951-954. doi: 10.3201/eid2505.180904. PMID 31002058